# Investigating Medical Research Trends in Osteoarthritis Clinical Trials: Analyzing Factors Impacting Patient Involvement

Consent Form for the Observational Clinical Study Conducted by Power Clinical Trial

Date: March 30, 2023

Detailed Overview and Consent Form for Our Observational Clinical Study

Welcome to our observational clinical study. The purpose of this study is to investigate the factors affecting clinical trial participation rates in patients with osteoarthritis. By completing questionnaires and participating in follow-up calls, we aim to understand why patients choose to enroll, remain, or withdraw from clinical trials.

We want to ensure that you have all the necessary information before deciding to participate in our research project. Your consent is required for participation, but you are under no obligation to do so and may withdraw at any time. The primary procedures of this observational clinical study have been designed to minimize any risks to participants, and as an observational study, there may not be any direct medical benefits.

However, the data collected can be used to identify ways to improve clinical trial participation rates and ultimately benefit patients with osteoarthritis. By participating in this study, you have the opportunity to contribute to the advancement of medical research and the improvement of clinical trial practices.

The findings of this study will provide valuable insights into the factors affecting clinical trial participation rates. This information can be used to improve recruitment strategies and patient engagement in clinical trials, ultimately benefiting osteoarthritis patients.

However, we want to emphasize that participation is voluntary and declining to participate will not affect your rights or privileges.

We want to ensure that you are fully informed before making a decision about participation. We encourage you to review this consent form carefully and ask any questions you may have. It is recommended that you discuss the study with your family, friends, trusted advisors, and healthcare professionals to make an informed decision. Remember that your participation is entirely voluntary, and you have the right to withdraw at any time without consequences.

Please read the consent form carefully before signing. By signing, you confirm that you have read and understood the information provided and that you consent to participate in this study.

### The Significance of This Clinical Trial

Clinical trials play a critical role in the advancement of new treatments for osteoarthritis. However, clinical trial participation rates may not accurately represent the broader population, and underrepresented groups often have low participation rates. Therefore, this clinical trial seeks to understand the variables that influence a patient's decision to participate in osteoarthritis clinical trials.

Our aim is to identify the factors that influence underrepresented groups' low participation rates and develop strategies to increase their participation rates. By doing so, we can increase the effectiveness and relevance of future clinical trials and ultimately improve osteoarthritis patients' lives.

It is important to emphasize that participation in this clinical trial is entirely voluntary, and participants have the right to withdraw at any time without any consequences. The study's primary procedures involve answering questionnaires and making follow-up calls, with minimal risk to the participants. We encourage potential participants to carefully review the consent form and ask any questions they may have before deciding to participate.

# Clinical Trial Methodology

Our research team is conducting an observational clinical study to investigate the factors that influence osteoarthritis patients' participation in clinical trials. As a

participant in an interventional trial, you have been invited to join our study. We will use electronic medical record systems to identify potential participants who meet our study's criteria. If you choose to participate, our staff will provide you with a consent form to sign, and they will explain the study's objectives and your rights as a participant.

To gather information about patient experiences with clinical trials, participants will be asked to complete a questionnaire every two weeks and participate in phone or video interviews every three months. These questions will ask about your medical history, demographics, and reasons for enrolling, withdrawing, or completing the clinical trial. All information collected will be kept confidential and anonymous.

Our research team will use statistical methods to analyze the data collected and identify the factors that influence patient participation in clinical trials. The results of this study will be presented at conferences and published in scholarly journals, with the aim of improving patient recruitment and retention in future clinical studies for osteoarthritis Participation in this study is entirely voluntary, and you have the right to withdraw at any time without consequence.

#### Potential Risks and Benefits of the Clinical Trial

Before deciding to participate in an observational clinical research study for osteoarthritis, potential participants should be aware of the risks and benefits involved. Risks may include privacy violations, emotional distress, and potential negative outcomes from any procedures conducted during the trial. However, the study team will take steps to protect participants' privacy and well-being.

On the other hand, participating in the study can provide an opportunity to contribute to medical research and potentially improve future treatment options for osteoarthritis. Additionally, participants may receive expert care and attention throughout the study. It is essential to carefully consider the potential risks and benefits and discuss any concerns with the study team and healthcare provider before making a decision.

#### Discontinuation of the Clinical Trial

While participants in clinical studies have the right to withdraw their consent and stop their involvement in the study at any time, it is also possible for the researcher or sponsor to discontinue a participant's involvement in the study for various reasons. These reasons could be due to factors such as the study being suspended or

terminated, the withdrawal, suspension, or removal of funding, or if it is considered to be in the participant's best interests.

Furthermore, there are participant-related reasons why the study team may decide to discontinue a participant's involvement in the study. For instance, if a participant experiences a decline in their health status during the study, or if they become pregnant, the study team may stop their participation. Additionally, if a participant chooses not to continue with the research after being informed of any changes that may affect them, or if they fail to adhere to the study's protocols, their involvement may be terminated.

Participants should be aware that discontinuing their involvement in the study does not necessarily mean that they will be excluded from medical treatment or care. The study team will work with the participant and their healthcare provider to ensure that they receive appropriate follow-up care. It is important for participants to understand the reasons why their participation may be stopped and to discuss any concerns with the study team before making a decision to participate.

#### Our Osteoarthritis Clinical Trial vs Other Trials

While there are many clinical trials available for various medical conditions, it's important to understand the specific differences between osteoarthritis clinical trials and others.

Osteoarthritis trials may involve different interventions depending on the trial's objectives. These interventions can have various risks and benefits, which will be explained in detail in the informed consent form. Potential participants should carefully read and understand this document before deciding whether to participate.

In addition, osteoarthritis trials may have unique eligibility criteria that may exclude certain patients based on factors such as age, stage of the condition, or previous treatments. This can make it challenging to find a suitable trial to participate in.

However, resources such as clinicaltrials.gov can provide a list of <u>osteoarthritis studies</u> you can check. There is also Power's reference page, which can help patients identify <u>osteoarthritis clinical trials</u> that meet their specific needs.

It's also essential to discuss any concerns or questions about osteoarthritis clinical trials with your doctor and the study team before deciding to participate. This will help ensure

that you fully understand the risks and benefits of participating in a particular trial and can make an informed decision about whether to enroll.

## **Explore More Clinical Trial Diversity Topics**

If you want to explore the subject of clinical trial diversity in greater depth, there are many online resources that can provide valuable information. Here are a couple of articles that you may find informative:

Clark, Luther T., Laurence Watkins, Ileana L. Piña, Mary Elmer, Ola Akinboboye, Millicent Gorham, Brenda Jamerson et al. "Increasing diversity in clinical trials: overcoming critical barriers." *Current problems in cardiology* 44, no. 5 (2019): 148-172.

Knepper, Todd C., and Howard L. McLeod. "When will clinical trials finally reflect diversity?." (2018): 157-159.

## Participant's Statement

In order to participate in the research study, it is essential that you sign this consent agreement, acknowledging and agreeing to the following:

Firstly, you have read and fully understood the informed consent form and are well-informed about the research project and its methods. Prior to making a decision, it is recommended that you discuss this information with others and seek additional perspectives.

Secondly, you have received satisfactory answers to all your queries about the research study, and you possess all the necessary information to make a well-informed decision about participating.

Thirdly, you have considered the advantages and risks of participating in the study, as well as any other options that may be available.

Fourthly, by voluntarily agreeing to participate in the study, you understand that this will not affect your legal rights in any way.

Lastly, you will be kept informed of any significant changes or updates to the study that may affect your decision to continue participating. This consent form has been made

| available to you, and you are signing. | encouraged to ask any question | ns you may have before |
|---|---|---|
| Participant's Signature | | |
| Name of Participant | Signature of Participant | <br>Date |
| Statement of Person Givi | ng Consent | |
| patient with a detailed descript had to the best of my ability. | vestigator of this study, certify the otion of the study and have addressed on the pation of the pat | ressed any questions they ent's decision to participate |
| Signature of the Person \ | Who Obtained the Consent | |
| Name | Signature | <br>Date |